CLINICAL TRIAL: NCT02183090
Title: Pharmacokinetics and Tolerability of a Single 15mg Meloxicam Dose Injected Intramuscularly Compared to a Single Oral 15 mg Meloxicam Tablet in Healthy Subjects. A Two-way Cross-over, Randomized, Open Study.
Brief Title: Pharmacokinetics and Tolerability of Meloxicam Injected Intramuscularly vs. Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.217
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Meloxicam

ARMS (2):
- Meloxicam ampoule (Experimental)
  Interventions: Drug: Meloxicam ampoule
- Meloxicam tablet (Active Comparator)
  Interventions: Drug: Meloxicam tablet

INTERVENTIONS:
Drug: Meloxicam ampoule
  Arms: Meloxicam ampoule
Drug: Meloxicam tablet
  Arms: Meloxicam tablet

SUMMARY:
Study to investigate the pharmacokinetics and tolerability of an intramuscular 15 mg meloxicam injection in comparison to the 15 mg oral tablet

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by results of screening
* Written informed consent in accordance with Good Clinical Practice and local legislation
* Age ≥ 18 and ≤ 50 years
* Broca > - 20% and < + 20%

Exclusion Criteria:

* Any findings of the medical examination (including laboratory, blood pressure, pulse rate and electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastro-intestinal tract ( except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* Hypersensitivity to meloxicam and/or non-steroidal antirheumatic agents
* Intake of drugs with a long half-life (>24 hours) (≤ 1 month prior to administration or during the trial)
* Use of any drugs which might influence the results of the trial (≤ 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (≤ 2 months prior to administration or during the trial)
* Smoker (>= 10 cigarettes or >= 3 cigars or >= 3 pipes/day)
* Inability to refrain from smoking on study days
* Known alcohol abuse
* Known drug abuse
* Blood donation (≤ 1 month prior to administration)
* Excessive physical activities (≤ 5 days prior to administration)
* History of hemorrhagic diatheses
* History of gastro-intestinal ulcer, perforation or bleeding
* History of bronchial asthma
* For female subjects:

  * Pregnancy
  * Positive pregnancy test
  * No adequate contraception e.g. sterilization, IUD (intrauterine device), oral contraceptives
  * Inability to maintain this adequate contraception during the whole study period
  * Lactation period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1998-11; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
AUC0-inf (total area under the plasma drug concentration-time curve) | up to 96 hours after drug administration
Cmax (Maximum drug plasma concentration) | up to 96 hours after drug administration
tmax (Time to achieve Cmax) | up to 96 hours after drug administration

SECONDARY OUTCOMES:
AUC0-t (Total area under the plasma drug concentration-time curve from time of administration to the time of the last quantifiable drug concentration) | up to 96 hours after drug administration
λz (apparent terminal elimination rate constant) | up to 96 hours after drug administration
t1/2 (apparent terminal elimination half-life) | up to 96 hours after drug administration
MRTtot (Mean residence time) | up to 96 hours after drug administration
CL/f (Apparent clearance of the analyte in plasma at steady state after extravascular multiple dose administration) | up to 96 hours after drug administration
Vz/f (Apparent volume of distribution during the terminal phase λz following extravascular administration) | up to 96 hours after drug administration
Change from baseline in vital signs (pulse rate, systolic and diastolic blood pressure) | Baseline, days 1-5 of each treatment period
Change from baseline in laboratory parameters | Baseline, days 1-2 and 5 of each treatment period
Number of patients with adverse events | up to 72 hours after day 5 of each treatment period
Tolerability of the intramuscular injection | before and 4 and 24 hours after application of study drug